CLINICAL TRIAL: NCT01874041
Title: Effect of Massage Therapy and Occlusal Splint Therapy on the Electromyographic Activity and Mandibular Range of Motion in Individuals With Temporomandibular Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, MSc, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1144-0809
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Temporomandibular Disorder
Keywords: Physical Therapy Modalities; Facial Pain; Orthodontic Appliances
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Massage; Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Massage group (Experimental): The massage group was submitted to three weekly 30-minute sessions of massage of the muscles of mastication over four consecutive weeks.
  Interventions: Other: Massage
- The occlusal splint group (Experimental): The occlusal splint group was submitted to treatment with an occlusal splint for four weeks.
  Interventions: Other: Occlusal splint
- Control group (No Intervention): The control group was not submitted to any form of intervention and was evaluated on two occasions, with a four-week interval between evaluations.

INTERVENTIONS:
Other: Massage
  Arms: Massage group
Other: Occlusal splint
  Arms: The occlusal splint group

SUMMARY:
The objectives of this study were to investigate the effects of massage therapy and occlusal splint therapy in the electromyographic activity and mandibular range of motion (ROM) in individuals with temporomandibular disorder (TMD) and compare the results with those obtained in a group of individuals without this disorder. Twenty-eight volunteers with TMD were randomly distributed into two groups, massage therapy and occlusal splint. Both treatments lasted 4 weeks. Fourteen individuals without TMD were consecutively allocated to the control group. The Fonseca's anamnestic index was used to characterize TMD and allocate the volunteers to either the intervention groups or control group. The electromyographic activity and Mandibular ROM was evaluated before and after treatment using a digital caliper. Two-way analysis of variance with the Bonferroni test was used for inter and intragroup comparisons (level of significance was set to 5%). Cohen's d was used to calculate the effect size.

ELIGIBILITY:
Inclusion Criteria:

* male and female volunteers
* aged 18 to 40 years

Exclusion Criteria:

* occurrence of missing teeth
* current use of orthodontic appliance
* history of systemic or joint disease
* current use of analgesic, anti-inflammatory agent or muscle relaxant and currently undergoing physical therapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mandibular range of motion | 1 year
  Mandibular range of motion(maximum active mouth opening, and right and left lateral excursion) was evaluated by a blinded examiner on two occasions (before and after treatment) using a digital caliper.

SECONDARY OUTCOMES:
Electromyographic activity | 1 year
  Electromyographic activity in the masseter and anterior temporal muscles. The right and left masseter and anterior temporal muscles were analyzed with surface EMG.

CONTACTS AND LOCATIONS:
Overall Officials: Cid Gomes, MSc, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gomes CA, El Hage Y, Amaral AP, Politti F, Biasotto-Gonzalez DA. Effects of massage therapy and occlusal splint therapy on electromyographic activity and the intensity of signs and symptoms in individuals with temporomandibular disorder and sleep bruxism: a randomized clinical trial. Chiropr Man Therap. 2014 Dec 15;22(1):43. doi: 10.1186/s12998-014-0043-6. eCollection 2014. PMID 25512839
- See also: Related Info — http://www.uninove.br